CLINICAL TRIAL: NCT02706600
Title: RESCUE-COPD 1 Randomised Trial of E-Health Platform Supported Care vs Usual Care After Exacerbation of COPD
Brief Title: Trial of E-Health Platform Supported Care vs Usual Care After Exacerbation of COPD
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: my mhealth Ltd (Industry)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHT/2015/039
Record Dates: First submitted 2015-07-30; First posted 2016-03-11 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Written Self Management (Other): The HealthQuest written self management plan was produced in 2013. It is a one page document which contains a written self management plan which can be individualised for the patient. It consists of a traffic light system to direct patients to the most appropriate action to take should their symptoms deteriorate.
  Interventions: Behavioral: Written Self management plan
- Online Self Management (Active Comparator): myCOPD is a system that can be accessed by patients using any device that can connect to the internet and can operate in any internet browser. It contains: Educational information, Inhaler technique videos explaining the correct technique required to use different inhaler devices licensed for use in people with COPD.
  Medication and symptom diaries. Appointment diary, pulmonary rehabilitation videos to promote and support exercises that can be done in the home.
  Oxygen Alert Card - Users can create their own oxygen alert card online A 5 Day local weather and pollution reports - Feed for reports come from the met office and DEFRA.
  A Self management plan, which consists of a traffic light system to direct patients to the most appropriate action to take should their symptoms deteriorate. The action plan is populated automatically with the information input by the patients.
  Interventions: Behavioral: myCOPD

INTERVENTIONS:
Behavioral: myCOPD — myCOPD is a system that can be accessed by patients using any device that can connect to the internet and can operate in any internet browser. It contains: Educational information, Inhaler technique videos explaining the correct technique required to use different inhaler devices licensed for use in people with COPD.
  Medication and symptom diaries. Appointment diary Bitesize pulmonary rehabilitation videos designed to promote and support exercises that can be done in a home setting.
  Oxygen Alert Card - Users can create their own oxygen alert card online A 5 Day local weather and pollution reports - Feed for reports come from the met office and DEFRA.
  A Self management plan, which consists of a traffic light system to direct patients to the most appropriate action to take should their symptoms deteriorate. The action plan is populated automatically with the information input by the patients.
  Arms: Online Self Management
Behavioral: Written Self management plan — The HealthQuest written self management plan was produced in 2013. It is a one page document which contains a written self management plan which can be individualised for the patient. It consists of a traffic light system to direct patients to the most appropriate action to take should their symptoms deteriorate.
  Arms: Written Self Management

SUMMARY:
There are currently 900,000 people in the UK with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD), The disease is progressive and often causes disabling symptoms such as chronic cough, breathlessness and reduced tolerance to exercise. National Institute for Health and Care Excellence (NICE) recommends that patients with COPD have a self management plan (SMP). The utilisation of SMP's has been shown to reduce healthcare utilisation, improve quality of life, and reduces the need for hospitalisation. Currently SMP's are delivered to patient in a paper format, myCOPD is a web based self management system which has been developed by Healthcare professional and patients encompasses the principles of Self management and offers a viable solution to a national recommendation.

The study will compare paper self management plans against the online version myCOPD. The study aims to recruit 60 patients with a diagnosis of COPD during their admission to hospital for an exacerbation or flare up of their COPD. Patients will be given an information sheet during their admission and prior to leaving hospital be asked if they wish to participate in the study. Patients will participate in the study for no less than two months and a maximum of three months. 30 patients will receive written self management and 30 will receive online self management. There will be a total of 4 visits for the duration of the study.

The screening visits will comprise of written or verbal consent, Demographics, Medical, exacerbation and healthcare utilisation history, Quality of Life questionnaires, inhaler technique assessment and delivery of either a written self management plan. The telephone visits will comprise of verbal consent and completion of the COPD Assessment Test. The End of Study visit will comprise of verbal consent, Demographics, Medical, exacerbation and healthcare utilisation history, Quality of Life questionnaires and assessment of inhaler technique.

DETAILED DESCRIPTION:
The study will compare paper self management plans against the online version myCOPD. The study aims to recruit 60 patients with a diagnosis of COPD during their admission to hospital for an exacerbation or flare up of their COPD. Patients will be given an information sheet during their admission and prior to leaving hospital be asked if they wish to participate in the study. Patients will participate in the study for no less than two months and a maximum of three months. 30 patients will receive written self management and 30 will receive online self management. There will be a total of 6 visits for the duration of the study.

Visit One - Screening Visit This visit will take place within two weeks of discharge from hospital in the participants home and comprise of written informed consent, Demographics, Medical, exacerbation and healthcare utilisation history, Quality of Life questionnaires, inhaler technique assessment This will be assessed using the critical errors list for each inhaler devices. Participants will also have their technique using each of their devices videoed. Those that fore fill inclusion and exclusion criteria will then be randomised in one of two groups, those receiving paper self management and those receiving online self management 'myCOPD'. For those receiving written self management The study nurse will complete with the participant a written self management plan. For those randomised to online self management they will be loan an android/iOS tablet computer and be given unique access codes and directed to the online 'How to tutorials .

Visit Two,Three - Telephone Visits There will be 2 telephone visits during the study and will comprise of verbal consent completion of the COPD Assessment Test and adverse event reporting.

Visit Four - End of Study Visit This visit will take place in the participants home and comprise of verbal consent, Demographics, Medical, exacerbation and healthcare utilisation history, Quality of Life questionnaires and assessment of inhaler technique. This will be assessed using the critical errors list for each inhaler devices and technique will be videoed. Participants will also be asked to complete a feedback questionnaire to evaluate user experience. Those allocated online will have their tablet computers collected by the study team and have a written self management plan delivered.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to complete all study procedures and give written informed consent.
2. A diagnosis of COPD defined as per the NICE COPD guidelines
3. Male or female volunteers aged 45+ admitted to hospital or the ambulatory care service with a primary diagnosis of acute exacerbation of COPD
4. Patients who are taking inhaled therapies for COPD
5. Current or ex-smokers with a pack year history of more than 10 years
6. Access to the internet and ability to operate web platform and or use written action plan

Exclusion Criteria:

1. Patients who have any another respiratory disease as their main complaint such as asthma, bronchiectasis, lung cancer, tuberculosis or any other significant respiratory disease.
2. Patients unable to read or use an Internet enabled device.
3. Patients with any uncontrolled medical condition which in the view of the principle investigator or their team would confound the impact of a COPD directed support tool.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 3 months
  This is a validated symptom scoring system used in COPD studies9 The CAT questionnaire contains eight questions and provides a reliable measure of the impact of COPD on health status. Patients read the two statements for each item, which describe the best and worst scenario, (e.g I never cough - I cough all the time), and decide where on the scale of 0-5 they fit. The maximum score is out of 40. The higher the CAT score the greater the impact of symptoms on their health status. Experts involved in the development of CAT suggest that any change of 2 or more in the patient's final score may indicate a clinically significant change. CAT will be recorded at the start prior to any intervention at visit one and 3 months post intervention at visit 4
Inhaler technique | 3 months
  As different inhaled medication devices require different techniques, each participant's inhaler technique will be assessed according to manufactures guidelines for each device and critical errors recorded. Their technique will be video recorded at visit one and visit two. Any changes to devices during the study will be recorded prior to starting any new treatment. Each participant's technique will be evaluated and the number of critical errors recorded for each device and a composite . Each device will have its own critical error list we have created based on manufactures guidelines. Participants technique will be videoed and assessed using a critical error list for each device by a Health care Professional. This assessment will take place at visit one prior to intervention and 3 months post intervention at visit 4. The difference in the number of errors for each device pre and post intervention will then be recorded.

SECONDARY OUTCOMES:
St Georges Respiratory Questionnaire (SGRQ) | 3 months
  The SGRQ questionnaire has 50 items with 76 weighted responses. It has good discriminative and evaluative properties and is responsive to therapeutic trials. It was developed and validated in both asthma and COPD and designed to measure the health impairment of patients with respiratory disease. We will be assessed at visit one prior to intervention and 3 months post intervention
modified MRC | 3 months
  The mMRC dyspnoea scale comprises five statements that describe almost the entire range of respiratory disability from none (Grade 0) to almost complete incapacity (Grade 4). It can be self-administered by asking subjects to choose a phrase that best describes their degree of breathlessness associated with activity. This will be assessed prior to and three months post intervention
Hospital Anxiety and Depression Score (HAD) | 3 months
  This clinical scale was developed in 1983 and is in common use in clinical and trial settings. It consists of 7 questions scored form 0-3 to create a score out of 21. It is easily administered and has been well validated for the assessment of patients with COPD. This will be assessed prior to and three months after intervention
Patient Activation Measure (PAM) | 3 months
  PAM is a tool used for measuring the level of patient engagement in their healthcare. It was designed to assess an individual's knowledge, skill and confidence for self-management. PAM is a 13-item scale that asks people about their beliefs, knowledge and confidence for engaging in a wide range of health behaviors and then assigns an activation score based on their responses to the 13-item scale. This will be assessed prior to and three months post intervention.
Work Productivity Activity Impairment (WPAI) | 3 months
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a well validated instrument to measure impairments in work and activities. The 6 questions relate to work absenteeism (hours missed work) Work presenteeism (impairment whilst working) and work productivity lost due to a health condition. This will be assessed prior to and three months post intervention
Veterans Specific Activity Questionnaire (VSAQ) | 3 months
  The VSAQ is validated Self administered questionnaire developed to estimate exercise capacity for the development of exercise prescription. The VSAQ consists of physical activities listed in progressive order according to their energy demand estimated by metabolic equivalents (METs). One MET is equal to resting oxygen consumption 3.5 ml/kg/min. Therefore, numbers of METs express the energy cost of physical activities as a multiple of the resting metabolic rate. This will be assessed prior to and three months post intervention
Exacerbation History | 3 months
  COPD exacerbation data will be collecting from their primary prescriber on their exacerbation history. The numbers of COPD exacerbations requiring oral antibiotics and/or oral steroids by the participants one year prior to starting the study will be recorded at visit one. If the participant has any exacerbations requiring oral antibiotics and/or steroids required during the period of the study this will be recorded at visit four.
Admission and readmission data | 3 months
  Admission and readmission data will be collected at visit 1 and visit 4 and verified by the GP patient records or other source data.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Green, Dr, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospital NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice KL, Dewan N, Bloomfield HE, Grill J, Schult TM, Nelson DB, Kumari S, Thomas M, Geist LJ, Beaner C, Caldwell M, Niewoehner DE. Disease management program for chronic obstructive pulmonary disease: a randomized controlled trial. Am J Respir Crit Care Med. 2010 Oct 1;182(7):890-6. doi: 10.1164/rccm.200910-1579OC. Epub 2010 Jan 14. PMID 20075385
- [Background] Bourbeau J, Bartlett SJ. Patient adherence in COPD. Thorax. 2008 Sep;63(9):831-8. doi: 10.1136/thx.2007.086041. PMID 18728206
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Jones PW, Adamek L, Nadeau G, Banik N. Comparisons of health status scores with MRC grades in COPD: implications for the GOLD 2011 classification. Eur Respir J. 2013 Sep;42(3):647-54. doi: 10.1183/09031936.00125612. Epub 2012 Dec 20. PMID 23258783
- [Result] Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupre A, Begin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Sante du Quebec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. Arch Intern Med. 2003 Mar 10;163(5):585-91. doi: 10.1001/archinte.163.5.585. PMID 12622605
- See also: NICE (2010). National guidelines for the management of COPD in adults in primary and secondary care. — https://www.nice.org.uk/guidance/cg101
- See also: Department of Health (2012) An Outcomes Strategy for COPD and Asthma: NHS Companion Document. — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/216531/dh_134001.pdf
- See also: Consultation on a strategy for services for chronic obstructive pulmonary disease (COPD) in England. — http://guidance.nice.org.uk/QS10
- See also: 4 National Institute for Health and Care Institute (2011) guidance.nice.org.uk — http://guidance.nice.org.uk/QS10